CLINICAL TRIAL: NCT01105065
Title: Effect of Brimonidine 0.15% on Retinal Blood Flow Autoregulation and Motion Detection in Patients With Normal Tension Glaucoma
Brief Title: Effect of Alphagan on Retinal Blood Flow Autoregulation and Motion Detection in Patients With Normal Pressure Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Louis Pasquale, MD, Director, Glaucoma Service and Associate Director Telemedicine, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-03-019 (75643)
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Glaucoma
Keywords: Normal Pressure Glaucoma
MeSH Terms: conditions — Glaucoma; Low Tension Glaucoma | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with RVD (Experimental): Patients who exhibited retinal vascular dysregulation at the initial visit. Intervention: brimonidine 0.15% three times per day for 8 weeks.
  Interventions: Drug: brimonidine 0.15%

INTERVENTIONS:
Drug: brimonidine 0.15% — One drop in each eye three times a day for 8 weeks.
  Other Names: Alphagan

SUMMARY:
The investigators have completed a study in which the investigators examined the response of the retinal circulation to changes in posture from sitting to lying down in patients with Normal Tension Glaucoma (NTG). This alteration in position produces changes in the local blood pressure at the entrance to the retinal vasculature. In a healthy retina, the vasculature adapts by dilating and constricting in order to maintain a steady blood flow rate. In an eye with NTG, this often does not occur. Upon analysis at the completion of the study , the investigators found that the patients who had been taking Alphagan (brimonidine) during the study did not exhibit the blood flow increases typical of NTG while lying down; instead, they maintained a steady blood flow rate as did the group of healthy control subjects. The investigators primary objective is to now demonstrate in a prospective study that Alphagan can restore retinal vascular autoregulatory function in patients with NTG who do not autoregulate. The investigators will also determine the effect of Alphagan treatment on the patients' ability to detect motion.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized clinical trial of POAG patients with a history of untreated IOP <22 mm Hg.

RETINAL VASCULAR AUTOREGULATION TESTING PROTOCOL:

At approximately 10 AM, we allowed subjects to sit for 15 minutes and then measured blood pressure and heart rate using a Keller Vital Signs Monitor (Keller Medical Specialties, Antioch, Illinois, USA). We measured seated IOP in both eyes using Goldmann applanation tonometry (Haag Streit USA, Mason, Ohio, USA) and 1 eye was dilated with tropicamide 1%. Baseline seated ocular perfusion pressure (OPP) was estimated using the standard formula: OPP=2/3 MAP - IOP, where MAP refers to mean arterial pressure. The factor of two-thirds adjusts for the decline in blood pressure between the brachial and ophthalmic artery with the subject sitting. We used the Canon CLBF 100 Laser Blood Flowmeter (Canon Inc, Tokyo, Japan) to measure baseline retinal arterial blood column diameter and centerline blood speed, which allows for automatic calculation of the blood flow rate. We chose a site along either the inferior temporal retinal artery or the superior temporal retinal artery adjacent to the optic disc for baseline measurements. Following the baseline measurements, the subjects assumed a posture typically used for face-on x-rays, reclining on their right side with their head supported by a foam wedge making a 24-degree angle from the horizontal. Subjects reclined for 30 minutes while brachial blood pressure and heart rate were automatically measured at 5-minute intervals. Laser Doppler blood flow measurements were obtained from the same arterial site that was used at baseline after approximately 15 and 30 minutes of reclining. Immediately following the 30-minute laser Doppler measurement, with the subject still reclining, we used the Perkins handheld applanation tonometry (Haag Streit USA) to remeasure IOP in the eye undergoing hemodynamic testing. In the reclined position, OPP was estimated using the following formula: OPPreclining = MAPreclining - IOPreclining, where MAPreclining is the mean brachial artery blood pressure measured in the left arm with the subject reclining on the right side. Subsequently, blood pressure, heart rate, and laser Doppler measurements were repeated after the subjects were reseated for 15 minutes.

Only patients who exhibited retinal vascular dysregulation continued in the study. We defined retinal vascular dysregulation based on the percentage change between the retinal blood flow measured while reclining for 30 minutes and the baseline seated measures. Previously, we found that healthy subjects exhibited a +6.5% +/- 12% blood flow change induced by 30 minutes of reclining. Thus, we defined the normal range of blood flow autoregulation as within 2 standard deviations of the mean percentage change found in this group, or -17.5% to +30.5%. Patients who exhibited retinal vascular dysregulation began an 8-week course of brimonidine 0.15% 3 times a day in both eyes. Subsequently, they returned at 10 AM and repeated the testing protocol described above. We obtained retinal hemodynamic measurements at the same retinal arterial site used during the initial visit. Each patient also underwent visual function testing in the eye that had hemodynamic studies both before and after 8-week treatment with brimonidine 0.15%.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will have no history of IOP > 24 mm Hg in either eye.
* All subjects will have open angles on gonioscopy with the filtering portion of the trabecular meshwork visible for 360° in both eyes.
* Previously or newly diagnosed patient are required to have HVFs that are reliable and show loss consistent with nerve fiber layer atrophy.
* Patients with glaucoma-like discs (CDR>0.7 in either eye) and normal/reliable visual fields who the PI has opted to observe without treatment will enter the study if they meet the other study criteria.
* In order to facilitate the retinal blood flow measurements, only subjects with refractive error within the range -10 to +10 diopters, no lens opacities greater than 1+ cortical spokes or 2+ nuclear sclerosis, and pupillary dilation of at least 6 mm following mydriasis will be included.

Exclusion Criteria:

* Patients with evidence of exfoliation or pigment dispersion syndrome in either eye.
* Patients with a cup/disc ratio > 0.8.
* Known history of allergy to brimonidine.
* Patients already on treatment with brimonidine will be excluded from the study.
* Diabetic retinopathy.
* History of ocular laser or incisional surgery in either eye.
* Use of systemic alpha-2 blockers.
* Pregnant or planning to become pregnant.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis R Pasquale, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feke GT, Bex PJ, Taylor CP, Rhee DJ, Turalba AV, Chen TC, Wand M, Pasquale LR. Effect of brimonidine on retinal vascular autoregulation and short-term visual function in normal tension glaucoma. Am J Ophthalmol. 2014 Jul;158(1):105-112.e1. doi: 10.1016/j.ajo.2014.03.015. Epub 2014 Apr 5. PMID 24709811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants enrolled but only 23 had retinal vascular dysregulation.
Groups:
- Patients With RVD: Patients who exhibited retinal vascular dysregulation at the initial visit. Intervention: brimonidine 0.15% three times per day for 8 weeks.
  Alphagan (brimonidine) 0.15%: One drop in each eye three times a day for 8 weeks.
Period: Overall Study
Arm/Group | Patients With RVD
Started | 23
Completed | 17
Not Completed | 6
Not completed — Adverse Event | 5
Not completed — Technical Problems | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With RVD
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] — age range: 35 years to 80 years
  years | 57.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Presence of Retinal Blood Flow Autoregulation
Description: We defined retinal vascular dysregulation based on the percentage change between the retinal blood flow measured while reclining for 30 minutes and the baseline seated measures. In a prior study, we found that healthy subjects exhibited a +6.5%±12% blood flow change induced by 30 minutes of reclining. Thus, we defined the normal range of blood flow autoregulation as within 2 standard deviations of the mean percentage change found in this group, or -17.5% to +30.5%.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Patients With RVD
Number analyzed (Participants) | 17
participants | 14
Statistical Analysis 1: Comparison: Patients With RVD; There would be no change in retinal vascular dysregulation after treatment with brimonidine; Test type: Superiority or Other; p < 0.0001, Chi-squared, Corrected

2. Secondary Outcome: Frequency Doubling Perimetry
Description: Frequency doubling perimetry was measured pre- and post treatment with brimonidine for 8 weeks.We used the full-threshold N-30 protocol to determine the visual field mean deviation, pattern standard deviation, and test duration in the eye that had hemodynamic testing. The results that are reported below are the mean deviation values recorded as part of the frequency doubling perimetry as these are the most significant.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: dB
Groups:
- RVD Patients Pre-brimonidine Treatment: Patients who exhibited retinal vascular dysregulation at the initial visit. The mean deviation frequency doubling perimetry values were measured in these patients before their treatment with brimonidine.
- RVD Patients Post-brimonidine Treatment: Patients who exhibited retinal vascular dysregulation at the initial visit. The mean deviation frequency doubling perimetry values were measured in these patients after their treatment with brimonidine.
Arm/Group | RVD Patients Pre-brimonidine Treatment | RVD Patients Post-brimonidine Treatment
Number analyzed (Participants) | 17 | 17
dB | -2.03 (3.50) | -2.77 (5.03)
Statistical Analysis 1: Comparison: RVD Patients Pre-brimonidine Treatment; A paired t-test was used to determine if their was a statistically significant difference between the mean deviation of the frequency doubling perimetry in the RVD patients pre and post brimonidine treatment; Test type: Superiority or Other; p = 0.28, paired t-test

ADVERSE EVENTS:
Arm/Group | Patients With RVD
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 5/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With RVD (N=23)
Allergic reaction (Eye disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No